CLINICAL TRIAL: NCT05578105
Title: Prevalence and Genetic Alternation of Autoimmune Polyglandular Syndrome Type II in Taiwan
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202112250RINC
Record Dates: First submitted 2022-10-10; First posted 2022-10-13 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Autoimmune Polyendocrine Syndrome Type II
MeSH Terms: conditions — Polyendocrinopathies, Autoimmune

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Autoimmune polyendocrine syndrome type II: patients with autoimmune polyendocrine syndrome type II
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — No intervention, only observation

SUMMARY:
Autoimmune polyendocrine syndrome (APS) is an autoimmune disease involving at least two endocrine organ. It is classified into type I and type II diseases. Among them, APS type II is more common. It is diagnosed when two of the three following diseases are diagnosed in the same patient, including type 1 diabetes mellitus, autoimmune thyroid disease, and primary adrenal insufficiency. In this study, we will observe the epidemiology, clinical characteristics, and genetic variants of APS II in Taiwan.

ELIGIBILITY:
Inclusion Criteria:

* Patients visited NTUH during 2006-2021, and had at least two of the three diseases: type 1 DM, primary adrenal insufficiency, and autoimmune thyroid disease.

Exclusion Criteria:

* Patients aged less than 20 years old

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We study patients with autoimmune polyendocrine syndrome type II
Sampling Method: Non-Probability Sample
Enrollment: 650 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Rates of endocrine organs involved | 2022/1/1 ~ 2026/12/31
  We will observe the rate of each endocrine organ involved, including adrenal gland, thyroid, and pancreas

CONTACTS AND LOCATIONS:
Overall Officials: Shyang-Rong Shih, MD, PhD, Study Director — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No